CLINICAL TRIAL: NCT06914557
Title: Scrambler Therapy With Duloxetine-based Usual Care vs Duloxetine-based Usual Care for Chemotherapy-induced Peripheral Neuropathy: A Randomized Phase II Pilot Trial.
Brief Title: Scrambler Therapy With Duloxetine-based Usual Care vs Duloxetine-based Usual Care for Chemotherapy-induced Peripheral Neuropathy.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Principal Investigator, Marcin Chwistek, MD, PROFESSOR/MD, Fox Chase Cancer Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 23-1043
Record Dates: First submitted 2025-03-24; First posted 2025-04-06 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: CIPN - Chemotherapy-Induced Peripheral Neuropathy; Pain
Keywords: CIPN; neuropathy; Chemotherapy-Induced Peripheral Neuropathy; Duloxetine; Scrambler Therapy
MeSH Terms: conditions — Pain | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Intervention Model Description: The investigators propose a randomized wait-list control study comparing the effectiveness of Scrambler therapy with duloxetine to duloxetine-based usual care, which is the current standard for CIPN treatment. Wait-list control studies allow the control group to cross over to the intervention arm after the control period. These studies are commonly used in behavioral trials to ensure all participants have access to a potentially beneficial intervention. Wait-list control designs may also enhance accrual if the intervention is perceived as desirable by participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Duloxetine Group (Other): Patients will be treated with Duloxetine as per Specialized Outpatient Palliative Care SOPC standard neuropathy treatment protocol
  Interventions: Other: Questionnaire and Physical Exam
- Scrambler + Duloxetine (Active Comparator): Patients' pharmacological treatment of their CIPN (including the management of duloxetine and other co-analgesics) will follow SOPC standard neuropathy treatment protocol
  Interventions: Device: Scrambler Therapy; Other: Questionnaire and Physical Exam

INTERVENTIONS:
Device: Scrambler Therapy — Scrambler therapy will be administered by the staff of the Supportive Oncology and Palliative Care team who have been trained in Scrambler therapy and have extensive experience providing it to patients with neuropathic cancer-related pain. Patients who meet the study criteria will be treated daily, Monday through Friday, for up to 10 sessions. The treatment may be terminated sooner if a patient experiences complete pain relief or if it is ineffective after five sessions. Patients will be closely monitored during the treatment. The treatment is non-painful and not associated with any significant adverse effects.
  Other Names: Scrambler device therapy
  Arms: Scrambler + Duloxetine
Other: Questionnaire and Physical Exam — 15-minute-long questionnaires evaluating Pain and degree of pain.
  Other Names: EORTC QLQ-CIPN20; PDQ

SUMMARY:
The investigators hypothesize that Scrambler therapy with duloxetine, compared to duloxetine-based usual care, will result in greater improvement in CIPN as measured by the BPI-Short Form. In addition, the investigators will further assess pain using the EORTC CIPN-20 and determine whether Scrambler therapy results in improved levels of function as measured with the PDQ, and a decreased need for opioid medications.

Our primary objective is to investigate whether Scrambler therapy with duloxetine is superior to duloxetine-based usual care in achieving at least a 50% reduction in pain scores, when comparing the cross-sectionally measured "average" pain score at day 35 to the cross-sectionally measured "average" pain score at baseline.

DETAILED DESCRIPTION:
Chemotherapy-induced peripheral neuropathy (CIPN) is a frequently experienced and often persistent side effect of many commonly utilized chemotherapy regimens. This list of agents includes platinum agents, taxanes, vinca alkaloids, and bortezomib. The estimated incidence of this toxicity, according to some sources, can be as high as 68.1% (95% CI: 57.7-78.4%) among patients with exposure to antineoplastic agents commonly known to cause neuropathy. Chemotherapy-induced peripheral neuropathy can be significant for many patients and can limit their ability to perform activities of daily living (ADLs). It is a frequent dose-limiting complication around which many oncologists must navigate.

While many agents have been studied to mitigate this complication, few have been shown to be effective or clinically significant. Duloxetine, perhaps the agent with the most evidence for use, showed a mean decrease in a patient's average pain score on the Brief Pain Inventory-Short Form (BPI-SF) of 1.06 versus 0.34 in the control arm (on an 11-point scale) (p = 0.003). Many other therapies have been proposed, such as gabapentin, tricyclic antidepressants (TCAs), cannabinoids, lidocaine, oral glutamine, cryotherapy, acupuncture, massage, and exercise-each with varying degrees of effectiveness. Despite these numerous therapies, duloxetine is the current standard of care for treating neuropathic pain, as evidenced by its inclusion in the National Comprehensive Cancer Network guidelines for the management of adult cancer pain.

Scrambler therapy is a novel treatment modality that has a growing body of evidence for neuropathic pain. It was originally developed by investigators at the University of Rome Tor Vergata following a series of preliminary clinical trials conducted from 1999 to 2006, involving 2,297 cases of various types of medication-resistant neuropathic pain. The machine uses five artificial neurons to transmit strings of "non-pain" signals based on a proprietary algorithm.

The investigators hypothesize that Scrambler therapy with duloxetine, compared to duloxetine-based usual care, will result in greater improvement in CIPN as measured by the BPI-Short Form. In addition, the investigators will further assess pain using the EORTC CIPN-20 and determine whether Scrambler therapy will result in improved levels of function as measured with the PDQ, and decreased need for opioid medications.

Our primary objective is to investigate whether Scrambler therapy with duloxetine is superior to duloxetine-based usual care in helping patients achieve at least a 50% reduction in pain scores when comparing the cross-sectionally measured "average" pain score (question 5 on the BPI) at day 35 to the score at baseline (day 1). The post-crossover outcomes will be included in the primary analysis. The first measurement on day 1 and the last measurement on day 35 will be used.

Secondary objectives:

Investigate the proportion of patients in each arm who achieve at least a 30% reduction in their cross-sectionally measured "average" pain score on the BPI from day 1 to day 35 and from day 1 to day 56.

Investigate the effectiveness of Scrambler therapy in groups stratified by receipt of neurotoxic cancer therapeutic agents prior to study enrollment, based on changes in "average pain score" on the BPI from day 1 to day 35 and day 1 to day 56.

Compare the change in average daily oral morphine requirements (i.e., dosage) by treatment arm from day 1 to day 35 and day 1 to day 56.

Investigate the proportion of patients in each arm who achieve at least a 50% improvement in PDQ score from day 1 to day 35 and day 1 to day 56.

Exploratory outcomes:

Examine whether the proportion of patients who achieve at least a 50% reduction in their pain scores at the end of day 35 after receiving both Scrambler therapy and duloxetine differs between those randomized to the Scrambler therapy arm versus those in the duloxetine-based usual care arm who decide to cross over to the Scrambler therapy arm.

Investigate the proportion of patients between arms with at least a 50% improvement in EORTC score from day 1 to day 35 and day 1 to day 56.

Investigate the percentage of patients in the Scrambler arm who maintain at least a 50% improvement in EORTC score at day 180.

ELIGIBILITY:
Inclusion Criteria:

1. Persons aged 18 years or older with cancer
2. Eastern Cooperative Oncology Group 0-2
3. At least a 4/10 average pain score prior to treatment
4. At least CTCAE version 5.0 grade 2 neuropathies.
5. Diagnosed CIPN based on chart review or oncologist diagnosis; will allow pre-existing diabetic neuropathy if symptoms are changing or worsening after chemotherapy.
6. Score of at least 4 on the Douleur-Neuropathique-en-4 Questions (DN4) questionnaire
7. Patients must have discontinued neurotoxic chemotherapy within the last 3 months with no additional therapy planned for the next 6 months after initiation of CIPN treatment.
8. Patients must be on duloxetine at least 30 mg po daily for at least 4 weeks prior to study initiation
9. Patients must be able to provide informed written consent.

Exclusion Criteria:

1. Children or adolescents
2. Pregnant or nursing patients
3. Presence of an implantable life supporting medical device or implantable drug delivery system
4. Patients with severe skin conditions preventing the proper application of electrodes
5. Patients currently on monoamine oxidase inhibitors MAOIs.
6. Patients currently receiving gabapentin who are unable to be weaned off for other medical reasons (ST requires tapering gabapentin).
7. Patients with a symptomatic neuropathy from any type of nerve compression (e.g. carpal tunnel or tarsal tunnel, radiculopathy, spinal stenosis, or brachial plexopathy)
8. Patients with leptomeningeal carcinomatosis- treated/stable brain metastases are allowed
9. Patients with severe depression, suicidal ideation, bipolar disease, alcohol abuse, a major eating disorder
10. Patients with uncontrolled epilepsy.
11. Patients who have previously attempted or undergone Scrambler therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
The difference in the proportion with a 50% reduction in pain scores when comparing the cross-sectionally measured "average" pain score at day 35 with the cross-sectionally measured "average" pain score at baseline (baseline = day 1). | At Day 35
  Investigate whether Scrambler therapy with duloxetine is superior to duloxetine alone in patient achievement of at least a 50% reduction in pain scores when comparing the cross-sectionally measured "average" pain score at day 35 to the cross-sectionally measured "average" pain score at baseline (baseline = day 1).

SECONDARY OUTCOMES:
Proportion of patients achieving ≥30% reduction in average pain score on BPI from baseline to day 35 and day 56: secondary analysis including wait-list control post-crossover outcomes. | At Day 35 & Day 56
  Investigate the proportion of patients between arms who achieve at least 30% reduction in their cross-sectionally measured "average" pain score on the BPI from baseline (day 1) to day 35 and from day 1 to day 56. The wait-list control outcomes post-crossover will be included in this secondary analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Chwistek, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
We are not planning on sharing individual participant data IPD with anyone else. We will publish the data once available.